CLINICAL TRIAL: NCT02759302
Title: MRI on Persons With Mutations in POMT2 Gene (LGMD2N)
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sofie Thurø Østergaard, Scholarship student, Rigshospitalet, Denmark
Other Study IDs: STO-POMT2
Record Dates: First submitted 2016-04-27; First posted 2016-05-03 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Limb-girdle Muscular Dystrophy
Keywords: MRI; LGMD; POMT2
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with LGMD2N: Five patients over 18 years old with genetically verified LGMD2N

SUMMARY:
POMT2 mutation is known to cause Walker Warburg Syndrome and Muscle-Brain-Eye syndrome. Recently it has been connected to limb girdle muscular dystrophy (LGMD), a disorder characterized by muscle weakness and atrophy of the proximal muscles of the shoulder and pelvic girdles. LGMD is classified based on its inheritance pattern and genetic cause into more than 31 different types. LGMD with POMT2 mutations is a new phenotype - type 2N. Very few patients with the LGMD2N phenotype has been reported. In this study, the investigators examine five new cases with the LGMD phenotype. The primary aim is to examine the muscle involvement using MRI.

ELIGIBILITY:
Inclusion Criteria:

* Persons with genetically verified mutations in POMT2

Exclusion Criteria:

* All contraindications for undergoing an MRI scan

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons diagnosed with LGMD2N in Denmark and France are invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
MRI scan for qualitative analysis of muscle involvement | One MRI scan per subject (exam lasts approximately 60 min.)
  The MRI protocol include T1-weighted brain and whole body examination. Four cross-sectional slices at shoulder, lumbar back, thigh and calf are chosen for qualitative analysis using the grading scale from 1 to 4 developed by Mercuri et al. (2007) to evaluate the involvement of muscles by looking at the fat infiltration.

SECONDARY OUTCOMES:
Muscle Biopsy | One muscle biopsy per subject (last approximately 15 min.)
  One muscle biopsy from each patient from the tibialis anterior muscle or the deltoid muscle will be analyzed for glycosylated α-dystroglycan, merosin and POMT2. (Concentration determined by standard biochemical analysis).
10 meter walk test | Exam last approximately 5 min
  Measurement of the time it takes to walk 10 meters.
Neurological examination and test of muscle strength | Exam last approximately 15 min.
  Muscle strength (in arms and legs) will be examined by the principal investigator based on the Medical Research Council (MRC) scale with values spanning from 5(=normal strength) to 1(=No contraction).
Questionnaires | Data will be collected once for patients with LGMD2N (exam last approximately 45 min.)
  Data will be collected using Minimal mental examination (MMSE)
Heart examination | Exam last approximately 45 min
  Echocardiography and Electrocardiogram (ECG).
Forced Vital Capacity (FVC) | Exam last approximately 15 min
  FVC is measured as the best of three attempts using a hand-held spirometer.
Electromyography (EMG) | Exam last approximately 30 min
  EMG is used for measuring nerve conducting velocity and neuromuscular activity with repetitive stimulation (3Hz).

CONTACTS AND LOCATIONS:
Overall Officials: Sofie T. Østergaard, Bsc., Principal Investigator — Copenhagen Neuromuscular Center, Department of Neurology, Rigshospitalet, Copenhagen University
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Ostergaard ST, Johnson K, Stojkovic T, Krag T, De Ridder W, De Jonghe P, Baets J, Claeys KG, Fernandez-Torron R, Phillips L, Topf A, Colomer J, Nafissi S, Jamal-Omidi S, Bouchet-Seraphin C, Leturcq F, MacArthur DG, Lek M, Xu L, Nelson I, Straub V, Vissing J. Limb girdle muscular dystrophy due to mutations in POMT2. J Neurol Neurosurg Psychiatry. 2018 May;89(5):506-512. doi: 10.1136/jnnp-2017-317018. Epub 2017 Nov 24. PMID 29175898